CLINICAL TRIAL: NCT05608161
Title: Correlation Between Peripheral Hearing Loss and Auditory Perception Impairment in Patients With Unilateral Sudden Deafness and Its Underlying Neural Mechanism
Brief Title: Speech Perception Impairment Follow Complete Recovery of Sudden Sensorineural Hearing Loss
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Ma Xin, chief physician, Peking University People's Hospital
Other Study IDs: SNH-SP-01
Record Dates: First submitted 2022-05-11; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Sudden Sensorineural Hearing Loss
Keywords: Unilateral sudden sensorineural hearing loss; information masking; energy masking; neural mechanisms
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Hearing Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with unilateral sudden deafness with complete recovery of peripheral hearing: The patients who recovered from sudden deafness underwent speech recognition rate tests under different masking conditions and different signal-to-noise ratio conditions within 2 weeks after complete recovery of peripheral hearing and were followed up 3 times at 1, 6, and 12 months after recovery. The test content is the same as the first time.
  Interventions: Diagnostic Test: speech in noise test
- Healthy control group: Age-, gender-, and educational-matched healthy controls were enrolled as healthy control group to test speech recognition rates under different masking conditions and different signal-to-noise ratio conditions.
  Interventions: Diagnostic Test: speech in noise test

INTERVENTIONS:
Diagnostic Test: speech in noise test — The noise masker was a stream of steady-state speech-spectrum noise, whose spectrum was representative of the average spectrum of target sentences. The speech masker was a 47-s loop of digitally combined continuous recordings for Chinese nonsense sentences. Patients from the idiopathic sudden sensorineural hearing loss (ISSNHL) group and control group were tested bilateral (left, right) speech-in-noise (SIN) perception of various signal-to-noise ratios (SNRs) under speech and noise masking conditions. Each participant has to complete four consequent levels of SNRs (-12, -8, -4, 0 decibel (dB) for most of control group, -8, -4, 0, 4 dB for ISSNHL group). In addition, the benefits of spatial separation cues under these two types of masking were analyzed.

SUMMARY:
At present, few research on the auditory perception function and possible neural mechanisms of unilateral sudden hearing loss patients with complete or partial recovery of peripheral hearing.This project evaluate the speech perception function in noise of unilateral sudden hearing loss patients with with complete and partial hearing recovery by cognitive behavioral experiments, event-related potentials (ERPs) and functional magnetic resonance imaging (fMRI), and longitudinal follow-up to explore its underlying neural mechanisms.

DETAILED DESCRIPTION:
In clinical practice, many unilateral sudden hearing loss patients with complete and partial recovery of peripheral hearing still complain of hearing discomfort, especially difficulty in speech recognition in noisy environments. At present, there is still a lack of research on the auditory perception function and possible neural mechanisms of unilateral sudden hearing loss patients with complete or partial recovery of peripheral hearing. From the perspective of cognitive psychology, this project uses cognitive behavioral experiments, event-related potentials (ERPs) and functional magnetic resonance imaging (fMRI) to evaluate the reverberation environment of unilateral sudden hearing loss patients with complete and partial hearing recovery, and longitudinal follow-up to explore its underlying neural mechanisms. The investigators hope to understand the possible difficulties of binaural processing and auditory perception in patients with unilateral sudden deafness, and to explore the changes of central and cortical functions. This study not only has important guiding significance for the treatment and rehabilitation of patients with unilateral sudden deafness, but also expands the research group on auditory perception function and the psychological and neural mechanisms involved in binaural processing, which has important theoretical significance.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old;
* patients with unilateral idiopathic sudden sensorineural hearing loss (at least three adjacent frequencies of hearing loss ≥ 30 dB );
* the first onset;
* Contralateral hearing is normal; 5) Hearing is cured after treatment

Exclusion Criteria:

* Sudden deafness with possible definite etiology, such as Meniere's disease, large vestibular aqueduct syndrome, trauma, retrocochlear tumor, etc.;
* Severe underlying diseases, heart disease, blood disease, pregnancy, breastfeeding, etc.;
* Suffering from other central diseases that may affect speech perception disorders, such as Alzheimer's disease, etc.;
* Those who cannot cooperate with the whole study inspection;
* Those who do not agree to be enrolled or refuse to sign the informed consent form;
* Those who are using may affect the Medications or treatments for speech perception disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral sudden sensorineural hearing loss who was treated in the outpatient department of our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-11-10 (Estimated); Primary Completion 2023-05-10 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Noisy speech recognition rate | Change from Baseline Noisy speech recognition rate at admission，6 months, 12 months and 18 months after hearing recovery
  The proportion of subjects correctly identifying the target sentence under different masking conditions and different signal-to-noise ratio conditions.

IPD SHARING:
Plan to Share IPD: No